CLINICAL TRIAL: NCT00749125
Title: fMRI Studies of Emotional Circuitry in Major Depression
Brief Title: fMRI Studies of Emotional Brain Circuitry in People With Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R01MH064821-04 (NIH); R01MH064821 (NIH); 5R01 MH06482104; DATR A3-NSM
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Depression
Keywords: Emotional Circuitry; fMRI
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Lexapro (Experimental): The depressed participants in this arm will be given Lexapro.
  Interventions: Drug: Lexapro
- 2 Control (No Intervention): The nondepressed participants in this arm will not be given any intervention for depression.

INTERVENTIONS:
Drug: Lexapro — 10 mg by mouth once per day for first 2 weeks, with psychiatric re-evaluation every 2 weeks to determine if any change in dosage is required, with a maximum of 20 mg per day
  Other Names: Escitalopram
  Arms: 1 Lexapro

SUMMARY:
This study will examine activation of a brain circuit that regulates emotion in depressed patients before and after treatment to see which areas of the brain are involved in chronic depression.

DETAILED DESCRIPTION:
Major depressive disorder can be a recurrent problem for many people, interfering with their ability to function normally in day-to-day life. Although research shows that activation in certain brain areas corresponds to certain emotional functions, it is not well known which specific changes in brain functioning are related to or caused by depression. A proposed theory holds that depression is related to abnormal regulation of emotions and thoughts. This study will focus particularly on a brain circuit involved in emotional regulation, which includes the amygdala, the affective division of the anterior cingulate (ACad), and dorsolateral prefrontal cortex (DLPFC). The amygdala detects critical emotional information, especially threats; the ACad judges relevance of motivational cues, detects conflict, and regulates emotional responses; and the DLPFC has a critical role in supporting a wide range of cognitive control functions. This study will compare brain scans from people with and without depression to attempt to clarify which changes in brain functioning are related to depression.

Participation in this study will last 8 weeks. All participants will undergo initial screening in a telephone interview, then a diagnostic interview and brief physical examination. After passing through screening, participants will schedule a functional magnetic resonance imaging (fMRI) scan. The fMRI scan, lasting approximately 2 hours, will take pictures of both brain structure and brain functioning during different tasks. Also at this visit but outside the fMRI scanner, participants will be asked to complete an additional 2 hours of tasks on a computer. Depressed participants will then be given Lexapro, an approved drug for the treatment of depression. Participants taking Lexapro will go to scheduled doctor's visits after 2, 4, and 6 weeks of treatment to assess health, effectiveness of the drug, and side effects. On the eighth week, all participants will again undergo fMRI scanning and computer testing. At both the initial and follow-up fMRI study visits, images of brain function and anatomy will be recorded, heart rate will be monitored, and anxiety and arousal will be measured in the computer tests.

ELIGIBILITY:
Depressed:

Inclusion Criteria:

* Participant meets DSM-IV criteria for major depressive disorder
* Minimum score greater than 18 on Hamilton Depression Inventory
* Participant is right handed
* Participant speaks English

Exclusion Criteria:

* Significant limitations that would interfere with testing procedures, such as uncorrected visual or hearing loss
* MRI contraindications, such as foreign metallic implants or a pacemaker
* Known primary neurological disorders, including dementia, stroke, encephalopathy, Parkinson's disease, brain tumors, multiple sclerosis, or seizure disorder
* Severe or unstable medical illness, such as a heart attack within the past 3 months, end stage cancer, or conditions or drugs that may cause depression (like systemic steroids or uncorrected hypothyroidism)
* Currently at risk for suicide
* Known allergy or hypersensitivity to escitalopram

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2001-07; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette I. Sheline, MD, Principal Investigator — University of Pennsylvania

REFERENCES:
- [Background] Sheline YI. Neuroimaging studies of mood disorder effects on the brain. Biol Psychiatry. 2003 Aug 1;54(3):338-52. doi: 10.1016/s0006-3223(03)00347-0. PMID 12893109
- [Background] Fales CL, Barch DM, Rundle MM, Mintun MA, Mathews J, Snyder AZ, Sheline YI. Antidepressant treatment normalizes hypoactivity in dorsolateral prefrontal cortex during emotional interference processing in major depression. J Affect Disord. 2009 Jan;112(1-3):206-11. doi: 10.1016/j.jad.2008.04.027. Epub 2008 Jun 17. PMID 18559283
- [Background] Sheline YI, Price JL, Yan Z, Mintun MA. Resting-state functional MRI in depression unmasks increased connectivity between networks via the dorsal nexus. Proc Natl Acad Sci U S A. 2010 Jun 15;107(24):11020-5. doi: 10.1073/pnas.1000446107. Epub 2010 Jun 1. PMID 20534464
- [Result] Sheline YI, Barch DM, Donnelly JM, Ollinger JM, Snyder AZ, Mintun MA. Increased amygdala response to masked emotional faces in depressed subjects resolves with antidepressant treatment: an fMRI study. Biol Psychiatry. 2001 Nov 1;50(9):651-8. doi: 10.1016/s0006-3223(01)01263-x. PMID 11704071
- [Result] Fales CL, Barch DM, Rundle MM, Mintun MA, Snyder AZ, Cohen JD, Mathews J, Sheline YI. Altered emotional interference processing in affective and cognitive-control brain circuitry in major depression. Biol Psychiatry. 2008 Feb 15;63(4):377-84. doi: 10.1016/j.biopsych.2007.06.012. Epub 2007 Aug 24. PMID 17719567
- [Result] Sheline YI, Barch DM, Price JL, Rundle MM, Vaishnavi SN, Snyder AZ, Mintun MA, Wang S, Coalson RS, Raichle ME. The default mode network and self-referential processes in depression. Proc Natl Acad Sci U S A. 2009 Feb 10;106(6):1942-7. doi: 10.1073/pnas.0812686106. Epub 2009 Jan 26. PMID 19171889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2004-2009. Participants from Washington University in St. Louis.
Pre-assignment Details: 99 participants started the study and were assigned to either the depressed or control group.
Groups:
- Control Participants: The nondepressed participants in this arm will not be given any intervention for depression.
  At both the initial (baseline) and follow-up (8 weeks following baseline visit) study visits, images of brain function and anatomy will be recorded.
- Depressed Participants: Following completion of their baseline study visit, the depressed participants will be given 8 weeks of antidepressant treatment as an intervention for depression.
  At both the initial (baseline) and follow-up (post-intervention) study visits, images of brain function and anatomy will be recorded.
Period: Overall Study
Arm/Group | Control Participants | Depressed Participants
Started | 47 | 52
Completed | 36 | 34
Not Completed | 11 | 18

BASELINE CHARACTERISTICS:
Groups:
- 1 Lexapro: The depressed participants in this arm will be given Lexapro.
  Lexapro: 10 mg by mouth once per day for first 2 weeks, with psychiatric re-evaluation every 2 weeks to determine if any change in dosage is required, with a maximum of 20 mg per day.
  At both the initial and follow-up fMRI (functional magnetic resonance imaging) study visits, images of brain function and anatomy will be recorded.
- 2 Control: The nondepressed participants in this arm will not be given any intervention for depression.
  At both the initial and follow-up fMRI (functional magnetic resonance imaging) study visits, images of brain function and anatomy will be recorded.
- Total: Total of all reporting groups
Arm/Group | 1 Lexapro | 2 Control | Total
Number analyzed (Participants) | 52 | 47 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 47 | 99
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Nine of the 108 participants enrolled in the study either withdrew from the study or were withdrawn as no-shows prior to assignment to a group, and were not included in any analyses.
  years | 36.04 (9.605) | 32.15 (8.228) | 34.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 22 | 19 | 41
Region of Enrollment [Number; unit: participants]
  United States | 52 | 47 | 99

OUTCOME MEASURES:

1. Primary Outcome: Activations in Different Cortical Regions Caused by Emotionally Evocative Task
Description: MRI scans from 41 participants (23 depressed and 18 controls), including fMRI scans using an emotional distractor task, were analyzed for differences between groups in activation in a priori regions (amygdala and DLPFC), measured with BOLD signal, for two conditions of the task - attend fearful and ignore fearful, both at baseline and following 8 weeks of treatment for the depressed group. Voxel-wise comparisons (ANOVAs) were performed to determine differences in activations between groups within these regions. Positive values reflect a BOLD activation in that region; negative reflects a BOLD de-activation in that region. We expect more positive values (greater activation) in depressed participants at baseline than in controls during the attend fearful task, and more negative values (greater de-activation) in controls at baseline than depressed during the ignore fearful task. These differences were expected to lessen significantly following treatment in the depressed group.
Time Frame: baseline and week 8
Population: 23 patients with major depression were matched with 18 demographically similar healthy controls. Depressed subjects were treated with Lexapro 10 mg/day, initiated immediately following the first fMRI scan.
Measure: Mean (Standard Deviation); unit: Voxels
Arm/Group | 1 Lexapro | 2 Control
Number analyzed (Participants) | 23 | 18
Voxels
  Baseline - Amygdala - attend fear | -0.021 (0.128) | 0.084 (0.135)
  Baseline - Amygdala - ignore fear | 0.021 (0.190) | -0.030 (0.146)
  Baseline - DLPFC - attend fear | 0.072 (0.092) | -0.025 (0.132)
  Baseline - DLPFC - ignore fear | 0.063 (0.129) | 0.073 (0.086)
  Time 2 - Amygdala - attend fearful | -0.031 (0.264) | -0.032 (0.178)
  Time 2 - Amygdala - Ignore fearful | -0.031 (.214) | -0.041 (0.161)
  Time 2 - DLPFC - Attend fearful | 0.026 (0.134) | 0.075 (0.121)
  Time 2 - DLPFC - Ignore fearful | 0.091 (0.161) | 0.109 (0.123)

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events during their 8 week participation in the study.
Arm/Group | 1 Lexapro | 2 Control
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/48
Other Adverse Events (participants affected / at risk) | 0/51 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No